CLINICAL TRIAL: NCT01281371
Title: Clinical Devolution of a Medication Change at Patients With Mono- or Combination Therapy With Sitaxentan to a Regime Without Sitaxentan.
Brief Title: Observation Study of the Medication Switch at Patients Treated With Sitaxentan to a Regime Without Sitaxentan
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. med. Walter E. Haefeli, Department of Clinical Pharmacology and Pharmacoepidemiology
Other Study IDs: K344
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — only remaining blood of the security laboratory for analysis of plasma concentrations of drugs
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to the withdrawal of Thelin (Sitaxentan) in December 2010 all patients with pulmonary hypertension treated with Sitaxentan need to be switched to an alternative therapy. This study will observe in which way the change of medication - in the clinical routine, without exception in charge of the treating physician - affects clinical and laboratory parameters and patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary hypertension
* Treatment with Sitaxentan

Exclusion Criteria:

* Inability or unwillingness to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Sitaxentan
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter E. Haefeli, Prof. Dr. med., Principal Investigator — Department of Clinical Pharmacology and Pharmacoepidemiology
Locations (1):
- Department of Clinical Pharmacology and Pharmacoepidemiology, Medical department of the University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany